CLINICAL TRIAL: NCT05682781
Title: Effects of Oral Nutritional Supplement With Dietary Counseling in Community Dwelling Older Adults at Risk of Malnutrition
Brief Title: Nutrition Intervention in Older Adults at Risk of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BL64
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Counseling (Active Comparator)
  Interventions: Other: Dietary Counseling
- Dietary Counseling + Oral Nutritional Supplement (Experimental)
  Interventions: Dietary Supplement: Oral Nutritional Supplement; Other: Dietary Counseling

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement — Oral Nutritional Supplement
  Arms: Dietary Counseling + Oral Nutritional Supplement
Other: Dietary Counseling — Dietary Counseling

SUMMARY:
Thailand is one of the fastest aging countries and older adults are at greater risk of having inadequate nutrient intake and malnutrition (undernutrition). In the community setting, malnutrition has been linked to low muscle mass, sarcopenia, increased incidence of disability and functional impairments. The objective of this prospective, multicenter, randomized controlled, open-label, parallel-design study is to determine the effects of an oral nutritional supplement with dietary counseling on body weight, in comparison with dietary counseling alone, in community dwelling older adults at risk of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged ≥60 years at risk of undernutrition.
2. Community-dweller.
3. Participant is community ambulant.
4. Participant does not have any chronic disease(s) or has stable chronic disease(s) at study entry.
5. Participant voluntarily signed and dated on an IRB approved informed consent form (ICF) and provided authorization prior to study participation.
6. Participant is able to communicate and follow instructions.
7. Participant is able to consume food and beverages orally.
8. Participant is willing to refrain from taking non-study oral nutritional supplements.
9. Participant is able and willing to follow study procedures and record data in diary and complete forms or assessments as needed.

Exclusion Criteria:

1. Participant diagnosed with type 1 or type 2 diabetes.
2. Participant has active infectious disease.
3. Participant has been diagnosed with severe gastrointestinal disorders.
4. Participant has been diagnosed with advanced renal disease or end stage organ or pre-terminal diseases or acute myocardial infarction within the last 30 days from the baseline visit.
5. Participant has active malignancy within the last five years, or is in current treatment for malignancy.
6. Participant has any condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.
7. Participant is taking part in another study that has not been approved as a concomitant study.
8. Participant has disorder or other conditions, that may interfere with study product consumption or compliance with study protocol procedures.
9. Participant has been diagnosed or known to be allergic or intolerant to milk products.
10. Participant has continuous oral nutritional supplement usage for 30 days prior to the baseline visit.
11. Participant has been taking herbals, dietary supplements, or medications during the past 30 days prior to the baseline visit that could profoundly affect body weight or appetite.
12. Participant has clinically significant ascites, pleural effusion, edema, or dehydration

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 60 days
  Measured in kg

SECONDARY OUTCOMES:
Malnutrition risk | Baseline, Study Day 30 and Study Day 60
  Malnutrition Universal Screening Tool is a widely used screening tool for malnutrition. It classifies participants into one of three nutrition status categories: low risk/score = 0, medium risk/score = 1, and high risk/score ≥ 2. Minimum value = 0, Maximum value = 6. Higher score indicates worse outcome, i.e., increased risk of malnutrition.
Body mass index (BMI) | Baseline, Study Day 30 and Study Day 60
  Weight (kg)/Height (m)2
Mid-upper arm circumference | Baseline, Study Day 30 and Study Day 60
  Measured in cm
Change in body weight | Baseline and Study Day 30
  Measured in kg
Energy intake | Baseline, Study Day 30 and Study Day 60
  24-Hour Dietary Recall: Researcher-led interview on food and drink intake the previous day. Nutrient analysis will be performed using a dietary analysis program.
Nutrient intake | Baseline, Study Day 30 and Study Day 60
  24-Hour Dietary Recall: Researcher-led interview on food and drink intake the previous day. Nutrient analysis will be performed using a dietary analysis program.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyuan Liu, RDN, MPH, Study Chair — Abbott Nutrition Research & Development
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok
  - The Department of Internal Medicine, Faculty of Medicine, Thammasat University, Pathum Thani